CLINICAL TRIAL: NCT01306955
Title: The Efficacy of Intravenous Pulses of Methylprednisolone in the Treatment of Patients With Ocular Involvement in Behcet's Disease, a Double Blind Pilot Study
Brief Title: The Efficacy of Methylprednisolone in the Treatment of Patients With Ocular Involvement in Behcet's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Farhad Shahram, MD, Professor, Rheumatology Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11192
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Behcet's Disease
Keywords: retinal vasculitis; posterior uveitis; methylprednisolone
MeSH Terms: conditions — Behcet Syndrome; Retinal Vasculitis; Uveitis, Posterior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylprednisolone (Active Comparator): patients who received methylprednisolone
  Interventions: Drug: methylorednisolone
- dextrose water 5% (Placebo Comparator): patients who received dextrose water 5% as placebo
  Interventions: Other: dextrose water 5%

INTERVENTIONS:
Drug: methylorednisolone — intravenous infusion of 1000 mg methylprednisolone in 100cc D/w 5% on 3 consecutive days at beginning of treatment
  Arms: methylprednisolone
Other: dextrose water 5% — intravenous infusion of 100cc D/w 5% on 3 consecutive days at beginning of treatment
  Arms: dextrose water 5%

SUMMARY:
The goal of this study is to examine the efficacy of 1gram/day intravenous pulses of methylprednisolone on 3 consecutive days in Behcet's patients with ocular involvement. A total of 34 Behcet's patients referring to Behcet's clinic in Shariati hospital whose problem was confirmed with new international criteria of Behcet's disease (ICBD) will be randomly assigned into one of the two equal groups of intervention or control. Behcet's patients are those with ocular involvement who were under the same cytotoxic treatment with cyclophosphamide and azathioprine. For the patients in the intervention group, intravenous infusion of 1000 mg methylprednisolone in 100cc D/w 5% or 100cc D/w5% on 3 consecutive days will be added to treatment diet. Then treatment will begin with oral prednisolone, 0.5 mg/kg. After that, all the patients were followed up with no other therapeutic intervention by study group. The patients will be visited every 2 months by an ophthalmologist and study group for 6 months in 3 settings. To estimate the ocular inflammation of patients, we use visual acuity, retinal and ocular posterior chamber inflammation index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Behcet's disease according to international criteria
* New or relapse of retinal vasculitis who received any cytotoxic or glucocorticoid since 2 months ago
* New or relapse of severe posterior uveitis who are candidate for cyclophosphamide and azathioprine according to their physician

Exclusion Criteria:

* Not Signing the informed consent
* Visual acuity lower than 1/10 by Snellen chart
* Presence of infectious diseases such as TB
* Presence of diabetes mellitus, hypertension, heart disease, liver disease, renal disease, or edema
* Presence of other glucocorticoid consumption contraindications

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
OCULAR IBDDAM INDEX | 14 months
  Iranian Behcet's disease Dynamic Activity measurement
VISUAL ACUITY | 14
  Check visual acuity with snellen chart by ophthalmologist

SECONDARY OUTCOMES:
Inflammation in retin | 14
  Check inflammation in retin by ophthalmologist
Inflammation in posterior chamber | 14
  Check inflammation in posterior uvea by ophthalmologist
inflammation in anterior chamber | 14
  check inflammation in anterior chamber by ophthalmologist

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Shahram, Professor, Principal Investigator — Rheumatology Research Center, Tehran University of Medical Science
Locations (1):
- Rheumatology Research Center, Tehran University of Medical Science, Tehran, Iran